CLINICAL TRIAL: NCT03579758
Title: Perioperative Chemotherapy Prior To and After Reoperation for Incidental Gallbladder Cancer - An International, Randomized Phase III Trial
Brief Title: Chemotherapy Before & After Surgery in Patients With Resectable Gallbladder Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This trial will open as an NCTN trial.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Shishir Kumar Maithel, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00103908; NCI-2018-00816 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU4338-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Stage I Gallbladder Cancer AJCC v8; Stage II Gallbladder Cancer AJCC v8; Stage IIA Gallbladder Cancer AJCC v8; Stage IIB Gallbladder Cancer AJCC v8; Stage III Gallbladder Cancer AJCC v8; Stage IIIA Gallbladder Cancer AJCC v8; Stage IIIB Gallbladder Cancer AJCC v8
MeSH Terms: conditions — Gallbladder Neoplasms | interventions — Capecitabine; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (capecitabine) (Active Comparator): Participants undergo re-resection (including partial liver resection and portal lymph node dissection). Participants then receive capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine
- Arm II (chemotherapy, capecitabine) (Experimental): Participants receive cisplatin IV over 1 hour and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Within 10 weeks of chemotherapy, participants undergo re-resection (including partial liver resection and portal lymph node dissection). Participants then receive capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Cisplatin — Given IV
  Other Names: CDDP; Cis-diamminedichloridoplatinum; Cismaplat; Cisplatinum; Neoplatin; Platamin; Platinol
  Arms: Arm II (chemotherapy, capecitabine)
Drug: Gemcitabine — Given IV
  Other Names: dFdCyd; Gemcitabine hydrochloride; Gemzar
  Arms: Arm II (chemotherapy, capecitabine)

SUMMARY:
This phase III trial studies how well chemotherapy before and after surgery works in treating participants with gallbladder cancer that can be removed by surgery. Drugs used in chemotherapy, such as cisplatin, gemcitabine, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before and after surgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the difference in overall survival (OS) at 3 years for patients with incidental gallbladder cancer (IGBC) who receive neoadjuvant gemcitabine hydrochloride (gemcitabine) and cisplatin (gem/cis) prior to reoperation followed by adjuvant capecitabine compared to patients who receive only adjuvant capecitabine after reoperation.

SECONDARY OBJECTIVES:

I. To determine the difference in recurrence-free survival (RFS) at 1 year for patients with IGBC who receive perioperative chemotherapy prior to and after re-operation compared to patients who receive only adjuvant chemotherapy after reoperation.

II. To assess the clinical effect of perioperative chemotherapy compared to only adjuvant chemotherapy after reoperation on resectability among 3 cohorts: all enrolled patients, all patients who undergo staging laparoscopy, and all patients who undergo laparotomy.

III. To compare the incidence of residual disease at the time of re-resection between patients who receive perioperative chemotherapy and those who receive only adjuvant chemotherapy.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants undergo re-resection (including partial liver resection and portal lymph node dissection) after incidental diagnosis of gallbladder cancer. Participants then receive capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive cisplatin intravenously (IV) over 1 hour and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Within 10 weeks of chemotherapy, participants undergo re-resection (including partial liver resection and portal lymph node dissection). Participants then receive capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed T1b, T2 or T3 gallbladder cancer discovered incidentally at the time of or following routine cholecystectomy for presumed benign disease
* Resectable disease at the time of enrollment based on high-quality, preoperative, cross-sectional imaging of the chest, abdomen, and pelvis (C/A/P)
* Enrollment and randomization within 12 weeks of initial cholecystectomy
* High-quality cross-sectional imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) performed within 4 weeks prior to enrollment
* Able to give informed consent
* Able to adhere to study visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status of < 2
* Absolute neutrophil count ≥ 1500/mm³
* Platelet count ≥ 100,000/mm³

Exclusion Criteria:

* Patients with histologically-confirmed Tis, T1a, or T4 tumors
* Unresectable gallbladder cancer at the time of enrollment based on high-quality, preoperative, cross-sectional imaging of the C/A/P
* Unable to sign informed consent
* Serum creatinine > 1.5 x upper limit of normal or estimated creatinine clearance (CrCl) < 45 ml/min
* Serum total bilirubin > 1.5 x upper limit of normal
* Presence of active infection
* Pregnant and/or breastfeeding
* Known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years after study start
  Overall survival (OS) is defined as time from randomization to death from any cause.

SECONDARY OUTCOMES:
Recurrence-free survival | From surgery to first observed disease recurrence or death from any cause, assessed at 1 year
  Recurrence-free survival (RFS) at one year, defined as time from surgery to first observed disease recurrence or death from any cause, among only patients who undergo complete, curative-intent re-resection. Disease recurrence will be based on findings from surveillance cross-sectional imaging of the chest, abdomen, and pelvis (CT or MRI, and any other additional imaging necessary to confirm recurrence). Patients who do not undergo reoperation or re-resection, have incomplete resections (R2), or who have gross evidence of distant metastases and/or T4 disease will be excluded from the RFS analysis
Overall resectability rate | Up to 3 years after study start
  Overall resectability rate is defined as the proportion of patients who successfully undergo a re-resection versus all enrolled patients. Patients who do not undergo reoperation or re-resection, have incomplete resections (R2), or who have gross evidence of distant metastases and/or T4 disease will be considered as unresectable for resectability analyses.
Resectability rate at diagnostic laparoscopy | Up to 3 years after study start
  Resectability rate at diagnostic laparoscopy is defined as the proportion of patients who successfully undergo a re-resection versus all patients who undergo staging laparoscopy. Patients who do not undergo reoperation or re-resection, have incomplete resections (R2), or who have gross evidence of distant metastases and/or T4 disease will be considered as unresectable for resectability analyses.
Resectability rate at laparotomy | Up to 3 years after study start
  Resectability rate at laparotomy is defined as the proportion of patients who successfully undergo a re-resection versus all patients who undergo laparotomy. Patients who do not undergo reoperation or re-resection, have incomplete resections (R2), or who have gross evidence of distant metastases and/or T4 disease will be considered as unresectable for resectability analyses.
Incidence of residual disease after or at the time of re-resection | Up to 3 years after study start
  Incidence of residual disease after or at the time of re-resection is defined as the presence of either microscopic or gross malignancy based on pathologic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shishir K. Maithel, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Stanford Cancer Institute Palo Alto, Stanford, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No